CLINICAL TRIAL: NCT06497348
Title: Application of an Exercise Program Versus Exercise Plus Manual Therapy in the Treatment of Adhesive Capsulitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cecilia Sánchez Pérez, principal investigator of the study Application of an exercise program versus exercise plus manual therapy in the treatment of adhesive capsulitis., University of Alcala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10111999
Record Dates: First submitted 2024-06-17; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Capsulitis of Shoulder; Frozen Shoulder
Keywords: "adhesive capsulitis"; "frozen shoulder"; "manual therapy"; "therapeutic exercise"
MeSH Terms: conditions — Bursitis | interventions — Musculoskeletal Manipulations; Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: The evaluation of each group will be carried out in different rooms of the university, a team of 6 physiotherapists divided into two groups, where 3 will evaluate with knowledge of the pathology and the other 3 without knowledge of it.
  The experimental group will receive mobilization treatment and exercises, while the control group will receive only exercises. Weekly one-hour sessions will be held, from Monday to Friday, with two times available for each patient. The experimental group, treated by physiotherapists who know the pathology, will be applied Maitland mobilization techniques, focused on passive neural and joint mobilizations. Flexion-extension, abduction-adduction, and external and internal rotation movements will be performed.
  The control group, treated by physiotherapists who will blindly evaluate the patients, will only be prescribed exercises, the same as the experimental group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will receive mobilization treatment and exercises, while the control group will receive only exercises. Weekly one-hour sessions will be held, from Monday to Friday, with two times available for each patient. Changes in pain, mobility and functionality will be recorded in an Excel document to monitor progress.
  To the experimental group, treated by physiotherapists who know the pathology, Maitland mobilization techniques will be applied, focused on passive neural and joint mobilizations. Flexion-extension, abduction-adduction, and external and internal rotation movements will be performed.
  Interventions: Other: manual therapy and exercises (experimental group) or only exercises (control group) in people with frozen shoulder
- control group (Active Comparator): The control group, treated by physiotherapists who will blindly evaluate the patients, will only be prescribed exercises, the same as the experimental group.
  Interventions: Other: manual therapy and exercises (experimental group) or only exercises (control group) in people with frozen shoulder

INTERVENTIONS:
Other: manual therapy and exercises (experimental group) or only exercises (control group) in people with frozen shoulder — They will be divided into two groups, one experimental (they will be mobilized and given exercises to see whether or not they gain joint range in the different movements of flexion-extension, abduction-adduction and internal rotation-external rotation) and another control group ( The patients will be blindly evaluated and they will be given the same exercises as the experimental group)

SUMMARY:
The main objective is to evaluate whether a treatment program combining manual therapy (joint mobilization) and exercise is more effective in the treatment of adhesive capsulitis than an exercise program applied in isolation.

The researchers will compare both groups (experimental group and control group) using the different techniques.

During the sessions, mobility will be evaluated with a goniometer and data will be recorded to monitor progress, maintaining a confidential record of the data.

ELIGIBILITY:
Inclusion Criteria:

* men and women from 40 to 60 years old, whether or not they carry out physical activity
* intervention through therapeutic exercise and/or joint mobility.

Exclusion Criteria:

* children
* older people
* people with previous shoulder pathology
* people with cognitive impairment who cannot complete questionnaires
* treatment that does not include exercise or joint mobility
* treatment with machines.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
evaluation of the improvement of shoulder mobility in patients with adhesive capsulitis by performing by an exercise program, mobilization or boths techniques. | 3-4 months
  study and measure if there is improvement in adhesive capsulitis of the shoulder with the proposed exercise programs versus exercise plus manual therapy in 108 subjects, 54 subjects in each group and a descriptive analysis of the data will be carried out, examining the initial homogeneity between the groups. in terms of the variables age, sex, pain, range of motion and functionality. The Shoulder Pain and Disability Index (SPADI) questionnaire and the visual analogue scale (VAS) will be used to assess pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermeria y Fisioterapia de la Universidad de Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD, since patient data will be recorded along with informed consent, to which only patients and researchers will have access.